CLINICAL TRIAL: NCT03969654
Title: ROSA Total Knee Post Market Study: Prospective Multicenter U.S. Study of the ROSA Total Knee System
Brief Title: ROSA Robot Used in Total Knee Replacement Post Market Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMU2018-34K
Record Dates: First submitted 2019-05-29; First posted 2019-05-31 (Actual); Results first posted 2024-05-03 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Knee Pain; Chronic Osteoarthritis; Avascular Necrosis of the Femoral Condyle; Moderate Varus, Valgus or Flexion Deformities; Rheumatoid Arthritis
MeSH Terms: conditions — Genu Valgum; Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Robotic Assisted TKA (Active Comparator): Robotic Assisted TKA
  Interventions: Device: PERSONA Total Knee; Device: Vanguard Total Knee; Device: NexGen Total Knee
- Conventional TKA (Active Comparator): Conventional TKA
  Interventions: Device: PERSONA Total Knee; Device: Vanguard Total Knee; Device: NexGen Total Knee

INTERVENTIONS:
Device: PERSONA Total Knee — Primary Total Knee Arthroplasty
Device: Vanguard Total Knee — Primary Total Knee Arthroplasty
Device: NexGen Total Knee — Primary Total Knee Arthroplasty

SUMMARY:
This is a prospective, multicenter clinical study designed to facilitate the collection and evaluation of workflow efficiency, patient pain and function, and adverse event data. This clinical study will include Persona, NexGen, and Vanguard product families using the ROSA Total Knee Robotic System or conventional instrumentation. The primary objective of this study is to collect and compare clinical and surgical data using the commercially available ROSA Total Knee robotic instrumentation and conventional instrumentation.

DETAILED DESCRIPTION:
The primary objective of this study is to collect and compare clinical outcomes data using the commercially available ROSA Total Knee robotic instrumentation and conventional instrumentation.The assessments will include:Planned vs actual component positioning, workflow efficiency, patient safety based on incidence and frequency of adverse events, and clinical performance measured by overall pain and function, quality of life data, and radiographic parameters.

ELIGIBILITY:
Inclusion Criteria:

* Patient is a minimum of 18 years of age
* Independent of study participation, patient is a candidate for commercially available Persona, NexGen, and Vanguard knee components implanted in accordance with product labeling
* Patient has participated in this study-related Informed Consent process
* Patient is willing and able to provide written Informed Consent by signing and dating the IRB or EC approved Informed Consent form
* Patient is willing and able to complete scheduled study procedures and follow-up evaluations

Exclusion Criteria:

* Patient is currently participating in any other surgical intervention studies or pain management studies
* Patient has underwent contralateral UKA or TKA within the last 18 months
* Hip pathology with significant bone loss (e.g. avascular necrosis of the femoral head with collapse, severe dysplasia of the femoral head or the acetabulum)
* Hip pathology severely limiting range of motion (e.g. arthrodesis, severe contracture, chronic severe dislocation)
* Patient is pregnant or considered a member of a protected population (e.g., prisoner, mentally incompetent, etc.)
* Patient has previously received partial or total knee arthroplasty for the ipsilateral knee

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2023-09-22 (Actual); Study Completion 2023-09-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hillary Overholser, Study Director — Zimmer Biomet
Locations (5):
- United States (5):
  - Vail-Summit Orthopaedics, Vail, Colorado
  - Cornerstone Orthopedics & Sports Medicine, a division of Orthopedic Centers of Colorado, LLC, Westminster, Colorado
  - SIU School of Medicine, Springfield, Illinois
  - Henry Ford Health System, Detroit, Michigan
  - OrthoVirginia Chippenham, North Chesterfield, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A maximum of 300 subjects are to be competitively enrolled in this study across all sites; a maximum of 10 U.S sites will contribute, with participating sites each enrolling up to 75 implanted knees. Sites will enroll up to 45 patients using The ROSA Knee System and up to 30 patients using Conventional instrumentation using a consecutive and concurrent approach; total study enrollment into these arms is not to exceed 180 subjects and 120 subjects respectively.
Units Other Than Participants: Knees
Period: Overall Study
Arm/Group | Robotic Assisted TKA | Conventional TKA
Started | 133; 133 Knees | 48; 48 Knees
Completed | 133; 133 Knees | 48; 48 Knees
Not Completed | 0; 0 Knees | 0; 0 Knees

BASELINE CHARACTERISTICS:
Units Other Than Participants: Knees
Groups:
- Total: Total of all reporting groups
Arm/Group | Robotic Assisted TKA | Conventional TKA | Total
Number analyzed (Participants) | 133 | 48 | 181
Number analyzed (Knees) | 133 | 48 | 181
Age, Categorical [Count of Units; unit: Knees]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 41 | 15 | 56
  >=65 years | 92 | 33 | 125
Sex: Female, Male [Count of Units; unit: Knees]
  Female | 74 | 28 | 102
  Male | 59 | 20 | 79
Ethnicity (NIH/OMB) [Count of Units; unit: Knees]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 132 | 47 | 179
  Unknown or Not Reported | 0 | 0 | 0
Kellgren Lawrence [Count of Units; unit: Knees] — Population: The Kellgren-Lawrence grade was determined by a Principal Investigator review of the preop knee images for a baseline measurement. A Kellgren-Lawrence grading scale score of greater than or equal to, or less than 3 was used to determine the severity of the units; a score of 3 indicates multiple osteophytes, definite joint space narrowing, sclerosis, and possibly bone deformity. (Kellgren-Lawrence score scale: 0 being no joint space narrowing to 4 being severe joint space narrowing)
  Knees
    number analyzed (Participants) | 128 | 46 | 174
    number analyzed (Knees) | 128 | 46 | 174
    KL Grade ≥ 3 No | 29 | 10 | 39
    KL Grade ≥ 3 Yes | 99 | 36 | 135

OUTCOME MEASURES:

1. Primary Outcome: Clinical Performance
Description: EQ-5D Questionnaire: A questionnaire completed by the Patient and assesses his/her General Health Status. The EQ5D is used to derive a Quality of life index used for health economics considerations. The scale is from 0-1, 0 being dead and 1 being the best possible score.
Time Frame: Pre-op (Baseline), 6 weeks, 3 months, and 1 year
Population: Only subjects with valid EQ5D scores at the follow-up time points are included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Knee
Arm/Group | Robotic Assisted TKA | Conventional TKA
Number analyzed (Participants) | 133 | 48
Number analyzed (Knee) | 133 | 48
score on a scale
  Preop: number analyzed (Participants) | 132 | 48
  Preop: number analyzed (Knee) | 132 | 48
  Preop | .540 (.268) | .442 (.256)
  6 Week: number analyzed (Participants) | 124 | 44
  6 Week: number analyzed (Knee) | 124 | 44
  6 Week | .740 (.166) | .763 (.179)
  3 Month: number analyzed (Participants) | 120 | 42
  3 Month: number analyzed (Knee) | 120 | 42
  3 Month | .826 (.137) | .842 (.128)
  1 Year: number analyzed (Participants) | 95 | 35
  1 Year: number analyzed (Knee) | 95 | 35
  1 Year | .889 (.145) | .891 (.137)

2. Primary Outcome: Oxford
Description: Oxford Knee Score: The Oxford Knee Score is a patient completed 12-question metric to rate a patient's knee pain and function using an ordinal 0 - 4 point scale. The total score is obtained by calculating the sum of the 12 items. The minimum score is 0 (most severe) and the maximum score is 48 points (least severe).
Time Frame: Pre-op (Baseline), 6 weeks, 3 months, and 1 year
Population: Only subjects with valid Oxford scores at the follow-up time points are included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Knee
Arm/Group | Robotic Assisted TKA | Conventional TKA
Number analyzed (Participants) | 133 | 48
Number analyzed (Knee) | 133 | 48
score on a scale
  Preop: number analyzed (Participants) | 132 | 48
  Preop: number analyzed (Knee) | 132 | 48
  Preop | 24.6 (9.2) | 22.2 (8.2)
  6 Week: number analyzed (Participants) | 124 | 44
  6 Week: number analyzed (Knee) | 124 | 44
  6 Week | 32.0 (7.6) | 32.5 (6.8)
  3 Month: number analyzed (Participants) | 120 | 42
  3 Month: number analyzed (Knee) | 120 | 42
  3 Month | 38.2 (6.8) | 38.5 (6.9)
  1 Year: number analyzed (Participants) | 95 | 35
  1 Year: number analyzed (Knee) | 95 | 35
  1 Year | 42.4 (5.4) | 41.2 (5.8)

3. Primary Outcome: Post-Operative Pain & Satisfaction
Description: Post-Operative Pain & Satisfaction Survey. The scale range for the level of satisfaction ranges is very satisfied, satisfied, uncertain, and unsatisfied.
Time Frame: 6 weeks, 3 months, and 1 year
Population: Only subjects with Patient Satisfaction form at the follow-up time points are included in the analysis.
Measure: Count of Units; unit: Knee
Units Other Than Participants: Knee
Arm/Group | Robotic Assisted TKA | Conventional TKA
Number analyzed (Participants) | 124 | 44
Number analyzed (Knee) | 124 | 44
Knee
  6 Week: Very Satisfied | 80 | 32
  6 Week: Satisfied | 32 | 9
  6 Week: Uncertain | 12 | 2
  6 Week: Unsatisfied | 0 | 1
  3 Month: number analyzed (Participants) | 120 | 42
  3 Month: number analyzed (Knee) | 120 | 42
  3 Month: Very Satisfied | 89 | 34
  3 Month: Satisfied | 22 | 7
  3 Month: Uncertain | 9 | 1
  3 Month: Unsatisfied | 0 | 0
  1 Year: number analyzed (Participants) | 95 | 34
  1 Year: number analyzed (Knee) | 95 | 34
  1 Year: Very Satisfied | 77 | 23
  1 Year: Satisfied | 11 | 8
  1 Year: Uncertain | 6 | 3
  1 Year: Unsatisfied | 1 | 0

4. Primary Outcome: Total Range of Motion
Description: Total Range of Motion Change from Preop to 1 year. The scale includes the total range of motion (0 degrees of knee extension (fully straightened knee) and 135 degrees of knee flexion) from preop to 1-year postop
Time Frame: Pre-op (Baseline), 6 weeks, 3 months, and 1 year
Population: Only subjects with valid ROM scores at the follow-up time points are included in the analysis.
Measure: Mean (Standard Deviation); unit: degrees
Units Other Than Participants: Knee
Arm/Group | Robotic Assisted TKA | Conventional TKA
Number analyzed (Participants) | 133 | 48
Number analyzed (Knee) | 133 | 48
degrees
  Preop: number analyzed (Participants) | 132 | 48
  Preop: number analyzed (Knee) | 132 | 48
  Preop | 121.0 (13.9) | 115.7 (16.2)
  6 Week: number analyzed (Participants) | 124 | 44
  6 Week: number analyzed (Knee) | 124 | 44
  6 Week | 114.5 (12.9) | 111.4 (11.1)
  3 Month: number analyzed (Participants) | 121 | 42
  3 Month: number analyzed (Knee) | 121 | 42
  3 Month | 121.1 (11.0) | 120.7 (9.7)
  1 Year: number analyzed (Participants) | 94 | 36
  1 Year: number analyzed (Knee) | 94 | 36
  1 Year | 122.7 (9.5) | 120.4 (10.8)

ADVERSE EVENTS:
Time Frame: All adverse events reported throughout each subject's length of participation in the study are included. Length of participation is defined as the implantation date through the date of study closure or the date of subject withdrawal for an average of 1 year.
Description: Subjects are counted only once in each category, even if they experienced more than one adverse event in the specific category.
Arm/Group | Robotic Assisted TKA | Conventional TKA
All-Cause Mortality (participants affected / at risk) | 0/133 | 0/48
Serious Adverse Events (participants affected / at risk) | 7/133 | 1/48
Other Adverse Events (participants affected / at risk) | 52/133 | 20/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Robotic Assisted TKA (N=133) | Conventional TKA (N=48)
Transverse Femur Fracture at site of ROSA pins (Surgical and medical procedures) | 1 (1) | 0 (0)
Patient seen for 2nd opinion at another orthopaedic provider. Diagnosed with tibial Loosening (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Stiffness/Limited Motion due to missing PT; Patient underwent open lysis of adhesions and poly swap. (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Patellar Periprosthetic Fracture (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Anemia and Melena (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Calf Pain/Possible DVT (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Robotic Assisted TKA (N=133) | Conventional TKA (N=48)
Hypotension (Cardiac disorders) | 1 (1) | 1 (1)
Hypertension (Cardiac disorders) | 0 (0) | 1 (1)
Contralateral Knee Replacement (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3)
Inability to eat/full/nausea/vomiting/diarrhea (Gastrointestinal disorders) | 1 (1) | 3 (3)
Urinary tract infection/unable to void (Renal and urinary disorders) | 2 (2) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Infection (non-knee) (Infections and infestations) | 1 (1) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Hip/DJD (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Nonunion Femur Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lumbar Stenosis/Degenerative Disc/Facet Disease (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Plantar Fascitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Contralateral Knee Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Right Frontal Ischemic Infarct (Nervous system disorders) | 2 (2) | 0 (0)
Neuro not intact to Left foot and ankle unable to Dorsiflex (Nervous system disorders) | 1 (1) | 0 (0)
Lytic Lesions in Thoracic Spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Amelanotic Melanoma Right Upper Arm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Possible DVT (Vascular disorders) | 1 (1) | 0 (0)
Nasal Bleeding (Vascular disorders) | 1 (1) | 0 (0)
Pulmonary Embolism (Vascular disorders) | 2 (2) | 0 (0)
Mild Crepitus (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Stiffness/Limited ROM (Musculoskeletal and connective tissue disorders) | 10 (10) | 2 (2)
Traumatic Injury/Twisting (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Superficial Infection of Incision (Infections and infestations) | 1 (1) | 0 (0)
Irritation of the distal aspect of Incision (Infections and infestations) | 1 (1) | 0 (0)
Severe Swelling of the surgical knee following surgery (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Trauma/Fall (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Periprosthetic Joint Infection (Infections and infestations) | 2 (2) | 0 (0)
Dermatitis/allergic reaction (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Arthritis Increased (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dizzy/Nausea from medication (Surgical and medical procedures) | 1 (1) | 0 (0)
Wound Dehiscence Left Ankle (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Stress Reaction at Femoral Pin Sites (Surgical and medical procedures) | 1 (1) | 0 (0)
Patella Dislocation (Surgical and medical procedures) | 0 (0) | 1 (1)
Skyline Patella Lateral Tilt and Erosion of Non-Resurfaced Patella (Surgical and medical procedures) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-02): https://cdn.clinicaltrials.gov/large-docs/54/NCT03969654/Prot_SAP_000.pdf